CLINICAL TRIAL: NCT05494190
Title: The Management of Metastatic Neck Nodes in N2/3 Hypopharyngeal Squamous Cell Carcinoma: A Multi-center Randomized Controlled Prospective Study
Brief Title: The Management of Metastatic Neck Nodes in N2/3 Hypopharyngeal Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Harbin Medical University Third Affiliated Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhang, Principal Investigator, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EENTHN0706
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypopharyngeal Carcinoma
Keywords: Metastatic Neck Nodes; Induction Chemotherapy; Neck Dissection
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine; Chemoradiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Induction chemotherapy group (Experimental): Patients initially receive induction chemotherapy consisting of docetaxel, cisplatin and capecitabine (TPC), q3w, 2-3 cycles in total.
  Patients with regional response of complete reaction (CR)/partial reaction (PR)≥50% after induction chemotherapy then receive concomitant chemoradiotherapy for both the primary and regional sites.
  Patients with regional response of PR<50%/stable disease (SD)/progressive disease (PD) after induction chemotherapy then receive surgery for both the primary and regional sites and postoperative concomitant chemoradiotherapy.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Capecitabine; Radiation: Concomitant chemoradiotherapy; Procedure: Surgery
- Surgery group (Active Comparator): Patients initially receive surgery for both the primary and regional sites and postoperative concomitant chemoradiotherapy.
  Interventions: Radiation: Concomitant chemoradiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Docetaxel — 60 mg/m2 i.v. day 1
  Arms: Induction chemotherapy group
Drug: Cisplatin — 60 mg/m2 i.v. day 1-3
  Arms: Induction chemotherapy group
Drug: Capecitabine — 750 mg/m2 po bid day 1-14
  Arms: Induction chemotherapy group
Radiation: Concomitant chemoradiotherapy — Radiotherapy: using intensity-modulated radiation therapy (IMRT)
  Gross tumor volume (GTV) for primary tumor: 66-70 Gy in total, 2.0~2.2 Gy per day, 5 days per week
  Clinical target volume (CTV) for lesions closely related to the primary lesion and metastatic lymph nodes: 65~70 Gy in total, 1.7~2.0 Gy per day, 5 days per week
  Prophylactic irradiation for sites of suspected subclinical spread: 50~60 Gy in total, 1.7~2.0 Gy per day, 5 days per week
  Concurrent chemotherapy: cisplatin 80 mg/m2 on days 1-3 every 3 weeks.
Procedure: Surgery — Neck dissection and primary tumor resection

SUMMARY:
This is a multi-center, multidisciplinary, open-label, randomized controlled prospective clinical study.

DETAILED DESCRIPTION:
Hypopharyngeal squamous cell carcinoma (HPSCC) is prone to have regional metastasis, which is an established negative prognostic factor. Especially for N2/3 patients whose metastatic neck nodes are bulky and have multiple or extracapsular spreads, their survival outcome is even worse. Therefore, it is vital for clinicians to select proper treatment and further improve the prognosis of N2/3 HPSCC patients. The aim of this randomized controlled prospective study is to explore the suitable treatment strategy of metastatic neck nodes in N2/3 HPSCC. This study will enroll a total of 111 HPSCC patients, who are clinically classified as T1/2 N2/3 M0 stage and initially treated with surgery (group 1) or induction chemotherapy (group 2). For patients with the regional response of PR<50%/SD/PD after induction chemotherapy, their following treatment will be surgery for both the primary and regional sites. For patients with the regional response of CR/PR≥50%, the following treatment will be concomitant chemoradiotherapy for both the primary and regional sites.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign a written informed consent document.
2. Age ≥ 18 and ≤ 75 years.
3. Male or female.
4. Karnofsky physical status (KPS): ≥ 80
5. Hepatic function, renal function and normal blood test. Hepatic function: Alanine aminotransferase (ALT) ≤ 2.5 upper limit of normal, Aspartate aminotransferase (AST) ≤ 2.5 upper limit of normal. Serum total bilirubin ≤ 1.5 upper limit of normal. Kidney function: Serum creatinine < upper limit of normal value and creatinine clearance rate > 60 ml/(min*1.73m2) (Cockcroft-Gault formula). Blood test: neutrophil (Neu) ≥ 1.5×109/L, platelet (PLT) ≥ 100×109/L, hemoglobin (HGB) ≥ 90 g/L.
6. Pathologically diagnosed with squamous cell carcinoma of the hypopharynx.
7. After clinical and radiographic evaluations, clinically classified as T1/2 N2/3 M0 stage according to American Joint Committee on Cancer (AJCC, eighth edition).
8. Resectable regional metastatic lesion (incompletely tumor- wrapped carotid vascular).
9. Assessable tumor lesions according to Response Evaluation Criteria in Solid Tumors (RECIST, Version 1.1).
10. Radical treatment intent.
11. Male patients with fertility and female patients with fertility and pregnancy risk must agree to use contraceptive methods throughout the study period, and continued until at least 6 months after the last dose of cisplatin. Female patients who do not have fertility (ie meet at least one of the following criteria): Have undergone hysterectomy and/or bilateral oophorectomy with archival records, medically confirmed ovarian function decline; In postmenopausal state. It is defined as: At least 12 months of continuous menstruation without other pathological or physiological reasons, and the status confirmed by serum follicle stimulating hormone (FSH) levels is consistent with postmenopausal status.
12. Good compliance.

Exclusion Criteria:

1. Distant metastatic disease
2. Have a history of other cancers or coinstantaneous second primary tumor
3. Previous treatment for the primary tumor, including radiotherapy, surgery except biopsy operation, chemotherapy, immunotherapy and biological targeted therapy.
4. Patients who have participated in other clinical trials within 1 month before the test.
5. Patients estimated to have poor tolerance to induction chemotherapy.
6. The investigator believes that it is inappropriate for individuals to participate in the trial: having, for example, severe acute or chronic medical conditions (including immune colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or mental illness (including recent time [within the past year] or active suicidal ideation or behavior).
7. Palliative treatment intent.
8. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 3 years
  The proportion of patients with disease progress or death due to any reasons.

SECONDARY OUTCOMES:
Overall survival rate | 3 years
  The proportion of dead patients due to any reasons.
Local control | 3 years
  The proportion of patients with local recurrence.
Regional control | 3 years
  The proportion of patients with regional recurrence.
Metastasis-free survival | 3 years
  The proportion of patients with distant metastasis.
Quality of life (UW-QOL V4.0) | 3 years
  Evaluated by University of Washington Quality of Life Questionnaire (UW-QOL) V4.0.
Adverse events | 3 years
  Evaluated by the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, PhD, Principal Investigator — Eye & ENT Hospital, Fudan University
Locations (3):
- China (3):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shandong Provincial ENT Hospital, Cheeloo College of Medicine, Shandong University, Jinan, Shandong
  - Eye & ENT Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No